CLINICAL TRIAL: NCT00592501
Title: A Phase II Study of Proton Radiotherapy With Chemotherapy for Nasopharyngeal Carcinoma
Brief Title: Proton Radiotherapy With Chemotherapy for Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Annie W. Chan, MD, Annie W. Chan, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-089
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: proton radiation; photon radiation; 5-FU; cisplatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Protons; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton/Photon Radiotherapy, Cisplatin, Fluorouracil (Experimental)
  Interventions: Radiation: Proton/Photon Radiotherapy; Drug: Cisplatin; Drug: Fluorouracil

INTERVENTIONS:
Radiation: Proton/Photon Radiotherapy — Given once a day, five days a week, for seven weeks.
Drug: Cisplatin — Given intravenously once every three weeks during radiation treatment, then once every four weeks for three cycles.
Drug: Fluorouracil — Given as continuous infusion over 4 days starting on the day cisplatin is received after radiation therapy.
  Other Names: 5-FU

SUMMARY:
Photon beam radiation is the standard type of radiation used to treat nasopharyngeal carcinoma. Photon beam radiation enters the body and passes through healthy tissue, encounters the tumor and leaves the body through healthy tissue. Proton beam radiation has been shown to have the same effect on tumors as photon beam radiation but it enters the body, passes through healthy tissue, and encounters the tumor but then stops. This means less healthy tissue is affected by proton beam treatment than by photon beam treatment. The purpose of this study is to determine the effectiveness of proton beam radiation in treating nasopharyngeal cancer and reducing the acute and long-term side effects from the treatment. This study will also test to see if the sparing of the healthy tissue can improve quality of life

DETAILED DESCRIPTION:
* Before beginning study treatment, participants will be asked to fill out a Quality of Life (QOL) questionnaires, a Speech Assessment, a ChemoSensory Questionnaire, a Patient Swallowing Diary, A Swallowing Study, Salivary Tests and a Trismus Assessment. Participants will need to go to the Massachusetts Eye and Ear Infirmary (MEEI) or Massachusetts General Hospital (MGH) for these tests.
* Radiation therapy will be given once a day, five days a week, for seven weeks. This will be given as outpatient care at the Northeast Proton Therapy Center (proton component) and Massachusetts General Hospital (photon component).
* During radiation treatments, participants will receive cisplatin intravenously once every three weeks. This three-week period is called a cycle of treatment.
* After the completion of radiation, participants will receive cisplatin intravenously once every 4 weeks along with fluorouracil as a continuous infusion over 4 days starting on the day cisplatin is given, for three cycles.
* Participants will have a physical exam and blood work drawn weekly to monitor their health.
* An MR/CT scan of the head and neck will be done 2 months after the radiation treatment.
* Follow-up visits will occur once every three months for 2 years, then once every 6 months during years 3-5, then annually. During these follow-up visits, participants will have the following tests and procedures: physical examination; blood work; chest CT scan and CT/MRI of the head and neck will be repeated once every 6 months during the first three years; swallow study; salivary study; QOL questionnaires; speech assessment; ChemoSensory Questionnaire; and Trismus Assessment.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven greater than or equal to T2b and/or node positive non-metastatic, squamous cell carcinoma of the nasopharynx, types WHO I-III.
* No head and neck surgery of the primary tumor or lymph nodes except incisional or excisional biopsies.
* Zubrod performance status 0-1 or Karnofsky 70 or above.
* All patients must undergo pre-treatment evaluation of tumor extent and tumor measurement.
* Nutritional and general physical condition must be considered compatible with the proposed chemoradiation treatment
* Patients must have adequate platelet and renal function as outlined in protocol.
* 18 years of age or above.
* No active alcohol addiction.
* Women of childbearing potential must have a negative pregnancy test.

Exclusion Criteria:

* Stage IVC or evidence of distant metastases
* Previous irradiation for head and neck tumor
* Patient is on other experimental therapeutic cancer treatment
* Other malignancy except non-melanoma skin cancer or carcinomas of head and neck origin and have been controlled for at least 5 years.
* Active untreated infection
* Major medical or psychiatric illness
* Prophylactic use of amifostine or pilocarpine
* Pregnant or breast feeding women
* Symptomatic peripheral neuropathy of grade 2 or greater by NCI CTCAE
* Symptomatic altered hearing > grade 2 by CTCAE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-10; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie W Chan, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period: 2006 and 2011 Location: Outpatient clinic at the Massachusetts General Hospital
Period: Overall Study
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
Started | 25
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Participant found to have metastatic disease after enrollment thus deemed ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 48 [32 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Toxicity
Description: Acute toxicities are side affects that occur during treatment and 90 days after completion.
Time Frame: 54 days of chemoradiation treatment and 90 days after completion, up to 144 days total
Measure: Count of Participants; unit: Participants
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
Number analyzed (Participants) | 23
Participants | 23

2. Primary Outcome: Participant Compliance Rate to Assigned Treatment Intervention
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
Number analyzed (Participants) | 23
percentage of participants
  Received at least 2 cycles of concurrent chemotherapy | 100
  Received at least 2 cycles of adjuvant chemotherapy | 75
  Received 3 cycles of concurrent chemotherapy | 83

3. Primary Outcome: Sialometry to Evaluate Xerostomia (Dry Mouth)
Description: Sialometry is a measure of saliva flow. The normal daily production of saliva varies between 0.5 and 1.5 liters. Stimulated saliva is produced in response to a mechanical, gustatory, olfactory, or pharmacological stimulus, contributing to around 40-50% of daily salivary production. In adults, normal total stimulated salivary flow ranges 1-3 mL/minute, low ranges 0.7-1.0 mL/minute, while hyposalivation is characterized by a stimulated salivary flow <0.7mL/minute.
Time Frame: Baseline and 2 years (24 months)
Population: The mean values below are for all analyzed participants.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
Number analyzed (Participants) | 23
milliliters
  Unstimatulated saliva at baseline | 1.89 (1.16)
  Unstimulated saliva at 24 months | 0.95 (0.57)

4. Primary Outcome: Penetration-aspiration Scale to Evaluate Swallowing Function
Description: The videofluoroscopic swallow study (VFSS) is the gold standard diagnostic tool to evaluate oropharyngeal dysphagia. The penetration-aspiration scale (PAS) is an 8-point scale used to grade the severity of penetration or aspiration observed in a videofluoroscopic swallow study. Aspiration is defined as the passing of the bolus below the true vocal folds, and penetration is when the bolus enters the airway but not below the true vocal folds. 1 is normal, no penetration or aspiration. 2-5 is penetration. 6-8 is aspiration.
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
Number analyzed (Participants) | 23
score on a scale
  Penetration-aspiration scale at baseline | 1.04 [1.00 to 2.00]
  Penetration-aspiration scale at 12 months after radiation therapy | 1.36 [1.00 to 5.00]

5. Primary Outcome: Serial Measurements of Maximal Inter-incisal Distance to Evaluate Trismus (Lockjaw)
Description: Serial measures of the changes of the maximal inter-incisal distance in the vertical opening, right lateral, and left lateral jaw movements are used to evaluate trismus (lockjaw). An average measurement of the three directional areas will be reported.
Time Frame: Baseline and 2 years
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
Number analyzed (Participants) | 23
millimeters
  Maximal inter-incisal distance at baseline | 51.4 (5.5)
  Maximal inter-incisal distance at 2 years | 43.8 (6.8)

6. Primary Outcome: ChemoSensory Questionnaire (CSQ) to Evaluate Smell and Taste Function
Description: The Chemosensory Questionnaire (CSQ) has four questions each on smell and taste. A minimum score of 4 and a maximum of 20 for the smell scale and taste scale are possible with a higher score indicating better function.
Time Frame: 2 years
Measure: Median (Standard Error); unit: score on a scale
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
Number analyzed (Participants) | 23
score on a scale
  Taste score post-treatment | 17 (1.05)
  Smell score post-treatment | 18 (1.06)

7. Primary Outcome: Number of Participants With Speech Problems Assessed by Head and Neck Health Status Assessment Inventory (HNHSAI)
Description: The Head and Neck Health Status Assessment Inventory (HNHSAI) is a descriptive outcome assessment consisting of 14 yes/no questions to measure number of participants with speech problems.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
Number analyzed (Participants) | 23
participants | 0

8. Primary Outcome: Health Related Quality-of-Life Outcomes Using Validated Quality-of-Life Instrument EORTC QLQ-C30
Description: General quality of life is measured with the European organization for research and treatment of cancer (EORTC) quality of life questionnaire (QLQ) EORTC QLQ-C30 (cancer 30). They are self-administered questionnaires. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for the global health status / QoL represents a high QoL.
Time Frame: 2 years
Measure: Median (Standard Deviation); unit: Global Health Status score on a scale
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
Number analyzed (Participants) | 23
Global Health Status score on a scale | 83 (20.9)

9. Primary Outcome: Health Related Quality-of-life Outcomes Using Validated Quality-of-life Instrument EORTC-QLQ-H&N
Description: General quality of life is measured with the European organization for research and treatment of cancer (EORTC) quality of life questionnaires (QLQ) for head and neck (H&N) (EORTC-QLQ-H&N). The head & neck cancer module incorporates seven multi-item scales that assess pain, swallowing, senses (taste and smell), speech, social eating, social contact, and sexuality. There are also eleven single items. All of the scales and single-item measures range in score from 0 to 100. For all items and symptom scales, high scores represent a high level of symptomatology/problems.
Time Frame: 2 years
Measure: Mean (Standard Error); unit: dry mouth score on a scale
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
Number analyzed (Participants) | 23
dry mouth score on a scale | 11.4 (3)

10. Secondary Outcome: Rate and Pattern of Locoregional Tumor Recurrence
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
Number analyzed (Participants) | 23
participants
  Local recurrence in high-dose region | 2
  Distant recurrence | 3

ADVERSE EVENTS:
Time Frame: Toxicity evaluation occurred during protocol therapy and 5+ years of follow-up.
Description: Adverse events were routinely collected through regular investigator assessment and regular laboratory testing.
Arm/Group | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil
All-Cause Mortality (participants affected / at risk) | 6/23
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil (N=23)
Blood/bone marrow (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton/Photon Radiotherapy, Cisplatin, Fluorouracil (N=23)
Constitutional Symptoms - Other (General disorders) | 1 (2) — "jittery"
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 2 (2) — Neutropenia
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1) — acid reflux
Renal failure (Renal and urinary disorders) | 2 (2) — acute renal failure
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2) — Alkaline phosphatase increased
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10)
ALT, SGPT (Metabolism and nutrition disorders) | 4 (7) — ALT increased
Neutrophils (Blood and lymphatic system disorders) | 6 (8) — ANC increased
Hemoglobin (Blood and lymphatic system disorders) | 13 (27) — Anemia (hemoglobin decreased)
Anorexia (Gastrointestinal disorders) | 21 (37)
Anxiety (Psychiatric disorders) | 11 (22)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection - lung (pneumonia) (Infections and infestations) | 4 (4)
AST, SGOT (Metabolism and nutrition disorders) | 2 (2) — AST increased
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 4 (4)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Infection - other (Infections and infestations) | 8 (13) — Candidiasis
Constitutional Symptoms - Other (General disorders) | 1 (1) — Carboplatin extravasation
Cardiac troponin T (cTnT) (Cardiac disorders) | 1 (1)
Infections - skin (cellulitis) (Infections and infestations) | 1 (1)
Rigors/chills (General disorders) | 4 (4)
CNS necrosis/cystic progression (Nervous system disorders) | 2 (2) — CNS necrosis
Confusion (Nervous system disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 12 (19)
Salivary gland changes/saliva (Gastrointestinal disorders) | 17 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dehydration (Gastrointestinal disorders) | 15 (25)
Mood alteration - Depression (Nervous system disorders) | 8 (10)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (4) — desquamation
Diarrhea (Gastrointestinal disorders) | 8 (10)
Dizziness (Nervous system disorders) | 12 (21)
Ophthalmoplegia/ diplopia (double vision) (Eye disorders) | 1 (1)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 20 (35)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) — DVT: left leg
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3 (4) — hoarseness
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 20 (33)
Neurology - other (Nervous system disorders) | 1 (1) — Dysosmia
Heartburn/dyspepsia (Gastrointestinal disorders) | 7 (7)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 22 (61)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lymphatics - other (General disorders) | 3 (3) — Edema unspecified
Edema: head and neck (General disorders) | 5 (5)
Edema: limb (General disorders) | 2 (3)
Hemorrhage, pulmonary/upper respiratory - nose (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Epistaxis
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 9 (11) — Erythema unspecified
Extrapyramidal/ involuntary movement/restlessness (Nervous system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 22 (63)
Febrile neutropenia (Infections and infestations) | 1 (1)
Fever (General disorders) | 5 (5)
Neuropathy: sensory (Nervous system disorders) | 7 (8)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1) — Soft palate defect
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6 (11)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Pain - head/headache (General disorders) | 9 (13)
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 15 (21) — Hearing loss
Hemorrhage/Bleeding - Other (Blood and lymphatic system disorders) | 1 (1) — Hemorrhage unspecified
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 13 (13)
Hypertension (Cardiac disorders) | 1 (1)
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 (4)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 4 (5)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 (8)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Cardiac disorders) | 3 (3)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ileus, GI (Gastrointestinal disorders) | 1 (1)
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1 (1) — "increased transaminase/LFT"
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) — c diff
Mucositis/stomatitis - oral cavity (Gastrointestinal disorders) | 17 (38) — thrush/oral mucositis
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 2 (2)
Insomnia (General disorders) | 6 (10)
Auditory/Ear - Other (Ear and labyrinth disorders) | 1 (1) — ear fullness
Tinnitus (Ear and labyrinth disorders) | 14 (29)
Pain - extremity-limb (General disorders) | 2 (4)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 9 (13) — leukocytes decreased
Lymphopenia (Blood and lymphatic system disorders) | 14 (20)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (2)
Memory impairment (Nervous system disorders) | 1 (1)
Constitutional Symptoms - Other (General disorders) | 19 (36) — mucositis unspecified
Mucositis/stomatitis - pharynx (Gastrointestinal disorders) | 15 (34)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 14 (25) — nasal congestion
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Nasal Stenosis
Nausea (Gastrointestinal disorders) | 21 (55)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 2 (2) — neck stiffness
Neurology - Other (Nervous system disorders) | 5 (5) — neuropathy unspecified
Apnea (Nervous system disorders) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 9 (18) — Odynophagia
Pain: oral-gums (General disorders) | 7 (15)
Infection - Middle ear (otitis media) (Infections and infestations) | 3 (3)
Pain NOS (General disorders) | 4 (7)
Pain - other (General disorders) | 3 (3) — pain at g-tube site
pain - anus (General disorders) | 1 (1)
pain - back (General disorders) | 3 (3)
pain - other (General disorders) | 1 (1) — ear pain unspecified
pain - face (General disorders) | 1 (1)
pain - eye (General disorders) | 1 (1)
pain - middle ear (General disorders) | 1 (1)
pain - neck (General disorders) | 1 (1)
pain - chest wall (General disorders) | 1 (1)
pain - oral cavity (General disorders) | 5 (9)
pain - throat/pharynx/larynx (General disorders) | 15 (22)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 (1) — Pancytopenia
neurology - other (Nervous system disorders) | 2 (2) — peripheral neuropathy unspecified
platelets (Blood and lymphatic system disorders) | 7 (9) — platelets decreased
infection - bronchus (Infections and infestations) | 1 (1)
pain - joint (General disorders) | 3 (3)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumomediastinum
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 11 (22)
weight loss (General disorders) | 22 (49)
Vasovagal episode (Cardiac disorders) | 1 (1)
Trismus (difficulty, restriction or pain when opening mouth) (Musculoskeletal and connective tissue disorders) | 9 (12)
infection - upper airway NOS (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 19 (33)
Syncope (fainting) (Nervous system disorders) | 2 (2)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 4 (5)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Sebaceous Cysts
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Rhinorrhea
Sweating (diaphoresis) (General disorders) | 2 (2)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1) — Soft palate fusion to post-oropharynx
Dermatology/Skin --Other (Skin and subcutaneous tissue disorders) | 2 (2) — Skin breakdown - lips
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 13 (28) — rash unspecified
Renal/Genitourinary - Other (Renal and urinary disorders) | 1 (1) — renal insufficiency
Infection - Other (Infections and infestations) | 1 (2) — ear infection unspecified
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — restless leg syndrome
Rash: dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 8 (14)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) — Thromboplebitis (left arm)
Constitutional Symptoms - Other (General disorders) | 1 (1) — thick mucus, unspecified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2011-06-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT00592501/Prot_SAP_000.pdf
  • Informed Consent Form (2012-02-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT00592501/ICF_001.pdf